CLINICAL TRIAL: NCT02587286
Title: Investigation of the Gather mHealth Platform on Diabetics' Behavior and Health Outcomes.
Brief Title: Gather mHealth India RCT for Behavior and Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gather Health India (Industry)
Collaborators: DHL Innovation Center, India (Other); Diabetes Action Centre (Other); M.V. Hospital for Diabetes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Gather mHealth 1
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: mHealth; Telemedicine; Randomized Controlled Trial; Glucose control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gather app (Experimental): Use of the Gather mHealth diabetes management system
  Interventions: Other: Gather app
- Control (No Intervention): Control group participants will be recruited from the same clinics and will also fit all study inclusion and exclusion criteria. Participants will be recommended to test their BG as per usual care in India. Providers will not contact control group participants between regular visits, though they will respond to queries directed at them in typical fashion.

INTERVENTIONS:
Other: Gather app — Participants in the intervention group will receive the Gather Health software free for the duration of the study. Their medication and BG testing goals will be entered into the system and they will receive automated reminders. Their data will be regularly reviewed by study staff and feedback provided.
  Arms: Gather app

SUMMARY:
The purpose of this trial is to explore the impact of the Gather Health diabetes management platform diabetics' health behaviors and health outcomes and how providers and diabetics interact with the Gather Health platform.

DETAILED DESCRIPTION:
The overall aim of the study is to estimate the impact of the Gather Health diabetes management platform on HbA1c, glycemic control, patient behavior, and physical and psychosocial measures. Additionally, this study will investigate patient and provider satisfaction with the platform.

Primary Objective:

Estimate the impact of the Gather Health diabetes management platform on HbA1c among diabetics in 3 cities in India.

Secondary Objective:

1. Estimate the impact of the Gather Health diabetes management platform on medication adherence, blood glucose (BG) control, body mass index (BMI), blood pressure (BP), and other behavior and health measures among diabetics in 3 cities in India.
2. Estimate patient and provider's satisfaction with the platform and the perceived usability and time spent on the platform
3. Generate ideas for future changes to the platform to make it more effective and user-friendly

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, diagnosis for > 6 months.
* Age 18-65, participants of either gender- males or females.
* HbA1c between 7.5% and 12.5% within last 6 months (inclusive).
* On stable diabetes therapy for >3 months prior to enrollment.
* Own an Android Smartphone.
* Participant willing to sign and date written Informed Consent Form to participate in the study.
* Willing to comply with the study schedule and procedures including randomization.

Exclusion Criteria:

* Previously used Gather Health
* Currently using an insulin pump or continuous glucose monitor.
* Pregnant or planning to become pregnant in the next 12 months.
* Severe hearing or visual impairment.
* Active substance, alcohol, or drug abuser (sober <1 year).
* Any psychiatric illness including psychosis or schizophrenia that will impair the patient's ability to complete the study or follow study protocol.
* Recent major surgery or planning to have major surgery
* Significant renal, hepatic, or other disease that may impair patient's ability to complete the study or follow study protocol
* Using glucocorticoids
* Patients who have received or are planning to receive an organ transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 6 months

SECONDARY OUTCOMES:
Change in HbA1c | 3 months

OTHER OUTCOMES:
BMI | 6 months
Blood pressure | 6 months
Waist Circumference | 6 Months
Fasting Blood Glucose | 6 Months
Lipids | 6 Months
Diabetes Self-care activities | 6 Months
Self-efficacy | 6 Months
  Stanford scale
Diabetes Knowledge | 6 Months
  Adaptation of RAND measure
Medication Adherence | 6 Months
  Visual Analog Scale
Blood Glucose Testing Adherence | 6 Months
  Visual Analog Scale
Treatment Satisfaction | 6 Months
  Adapted RAND measure
Diabetes Distress | 6 Months
  PAID-5
mHealth intervention satisfaction | 6 Months
  Investigator generated
BMI | 3 months
Blood pressure | 3 months
Waist Circumference | 3 months
Fasting Blood Glucose | 3 months
Lipids | 3 months
Diabetes Self-care activities | 3 months
Self-efficacy | 3 months
  Stanford Scale
Diabetes knowledge | 3 months
  Adapted RAND measure
Med Adherence | 3 months
  Visual Analog Scale
BG Testing Adherence | 3 months
  Visual Analog Scale
Treatment Satisfaction | 3 months
  Adapted RAND measure
Diabetes Distress | 3 months
  PAID-5
mHealth intervention satisfaction | 3 months
  Investigator generated

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Shah, MD, Principal Investigator — Diabetes Action Centre

IPD SHARING:
Plan to Share IPD: Yes
posted to clinicaltrials.gov

REFERENCES:
- [Derived] Kleinman NJ, Shah A, Shah S, Phatak S, Viswanathan V. Improved Medication Adherence and Frequency of Blood Glucose Self-Testing Using an m-Health Platform Versus Usual Care in a Multisite Randomized Clinical Trial Among People with Type 2 Diabetes in India. Telemed J E Health. 2017 Sep;23(9):733-740. doi: 10.1089/tmj.2016.0265. Epub 2017 Mar 6. PMID 28328396
- [Derived] Kleinman NJ, Shah A, Shah S, Phatak S, Viswanathan V. Impact of the Gather mHealth System on A1C: Primary Results of a Multisite Randomized Clinical Trial Among People With Type 2 Diabetes in India. Diabetes Care. 2016 Oct;39(10):e169-70. doi: 10.2337/dc16-0869. Epub 2016 Aug 4. No abstract available. PMID 27493133